CLINICAL TRIAL: NCT07158476
Title: Efficacy of Methylprednisolone for Pain Control After ACL Repair: A Randomized Controlled Trial
Brief Title: Efficacy of Methylprednisolone for Pain Control After ACL Repair
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Scott Kaar, MD, Professor, Orthopaedic Surgery, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 34336
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: ACL Surgery; Pain Management
Keywords: pain; opioids; orthopedic surgery
MeSH Terms: conditions — Agnosia; Pain | interventions — Meloxicam; Methylprednisolone; Gabapentin; Hydrocodone; Acetaminophen; Ketorolac; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medrol group (Active Comparator): Patients will receive Medrol dose pack, Meloxicam, Hydrocodone/Acetaminophen, and Gabapentin as pain regimen upon discharge from surgery.
  Interventions: Drug: Meloxicam 15 mg; Drug: Medrol 4 MG Oral Tablet Includes Medrol Dosepak; Drug: Gabapentin 300 mg; Drug: Hydrocodone 5Mg/Acetaminophen 325Mg Tab
- No Medrol group (Active Comparator): Patients will receive Ketorolac, Hydrocodone/Acetaminophen, and Gabapentin as pain regimen upon discharge from surgery.
  Interventions: Drug: Gabapentin 300 mg; Drug: Hydrocodone 5Mg/Acetaminophen 325Mg Tab; Drug: Ketorolac 10 Mg Oral Tablet

INTERVENTIONS:
Drug: Meloxicam 15 mg — PO once/day for 1 week
  Arms: Medrol group
Drug: Medrol 4 MG Oral Tablet Includes Medrol Dosepak — PO 6 day taper
  Arms: Medrol group
Drug: Gabapentin 300 mg — PO every 8 hours for 1 week
Drug: Hydrocodone 5Mg/Acetaminophen 325Mg Tab — PO 1-2 tabs every 4 hours as needed (total of 28 pills)
Drug: Ketorolac 10 Mg Oral Tablet — PO every 6 hours for 5 days
  Arms: No Medrol group

SUMMARY:
Opioids are commonly used after orthopedic surgery for pain control but have been shown to increase complications, surgeries, readmissions, and risk for opioid use disorder. The purpose of this study is to investigate the impact of adding a methylprednisolone taper to the pain regimen after ACL repair surgery to determine if this results in decreased postoperative pain and opioid use without increasing complications.

DETAILED DESCRIPTION:
The study is to include consecutive patients who undergo ACL repair by fellowship trained surgeons at a single institution with minimum 12 week follow up. All patients between the ages of 13-50 who are willing and able to provide informed consent will be included. Patients will be assessed preoperatively and then at 2 weeks, 6 weeks,12 weeks, and 1 year clinic visits, which is standard of care. The patient will fill out 2 questions on the MyCap app the day of surgery and for 14 days following surgery for pain scores and 15 days for amount of opioid pills consumed the day prior. Patient demographic, comorbidity, and surgical data will be collected from the medical record, including age, sex, BMI, smoking status, and diabetic status.

Patients will be randomized to the treatment or control group. The treatment group will receive the following pain regimen after surgery: Medrol dose pack, Meloxicam, Hydrocodone/Acetaminophen, and Gabapentin. The control group will be prescribed: Ketoralac, Hydrocodone/Acetaminophen, and Gabapentin. Pain reporting and opioid consumption will be assessed via the MyCap app for two weeks following surgery.

Patients will be followed at standard of care clinic appointments for 1 year. PROMs data will be collected at that time, in addition to any complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing ACL repair or ACL reconstruction with tendon autograft
* Age 13-50 years old
* Able to provide informed consent or parent/legal guardian is able for minors

Exclusion Criteria:

* Concurrent and significant injury to other bones or organs (Injury Severity Score of 4 or greater)
* Revision ACL reconstruction
* Concomitant additional ligament reconstruction or high tibial osteotomy
* A history of alcohol abuse, substance abuse or chronic opioid use (filled opioid medication ×2 within 6 months of the surgery)
* A history of renal failure (<60 mL/min/1.73 m2), liver dysfunction (child class, >B), severe heart disease (NYHA Class 4), diabetes, neurological or psychiatric diseases that may affect pain perception, and pre-existing immune suppression.
* A history or active peptic ulcer disease, gastrointestinal bleeding, or current use of anticoagulation.
* Patients currently taking oral or injectable glucocorticoids and those who have taken either within 1 month of the procedure.
* Patients who are currently pregnant.
* Patients who are unable to undergo the multimodal pain standardized protocol including those with comorbidities or medical allergies precluding the use of corticosteroids, gabapentin, hydrocodone, acetaminophen, ketorolac, and/or meloxicam.

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) pain scores | Post-op days 0-14, 2 weeks, 6 weeks, and 12 weeks
  Zero is equivalent to no pain and 10 indicates the worst possible pain

SECONDARY OUTCOMES:
Opioid consumption after surgery | 0-14 days postoperative
  Calculated using Morphine milligram equivalents (MME)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kaar, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No